CLINICAL TRIAL: NCT03077464
Title: Behaviorally Oriented Nutrition Education at a Russian Summer Camp: A Quasi-experimental Superiority Trial
Brief Title: Behaviorally Oriented Nutrition Education at a Russian Summer Camp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Responsible Party: Principal Investigator, Richard R. Rosenkranz, Associate Professor, Kansas State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KSU-CHE-FNDH-RussCamp
Record Dates: First submitted 2017-02-22; First posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Health Education; Healthy Eating; Health Knowledge, Attitudes, Practice
Keywords: nutrition education; Vegetables; Fruit
MeSH Terms: conditions — Health Education; Behavior

STUDY DESIGN:
Intervention Model Description: Non-randomized parallel group design, testing pretest to post-test changes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- behavioral nutrition education (Active Comparator): Set of curricular nutrition education modules, previously developed and based on Social Cognitive Theory, for the HOP'N After-School program, with additional materials from MyPlate. Materials were employed to increase healthy eating behavioral capability, self-efficacy, attitudes, and enjoyment. Topics included: 1) nutrition label literacy; 2) drinking water; 3) eating colors of the rainbow; 4) healthful snacks; 5) benefits of fruit and vegetable consumption; 6) moving more and sitting less; and 7) taking healthy habits home.
  Interventions: Behavioral: Behavioral nutrition education
- behavioral nutrition education plus skills (Experimental): Set of curricular nutrition education modules, previously developed and based on Social Cognitive Theory for the HOP'N After-School program, with additional materials from MyPlate. Materials were employed to increase healthy eating behavioral capability, self-efficacy, attitudes, and enjoyment. Topics included:1) nutrition label literacy;2) drinking water;3) eating colors of the rainbow;4) healthful snacks;5) benefits of fruit and vegetable consumption;6) moving more and sitting less;and 7) taking healthy habits home. Designed to differ from behavioral nutrition education condition by devoting at least 15 minutes of each session to an additional behavioral skills training component. The behavioral skills component was designed to bolster behavioral capability, healthy eating attitudes, self-efficacy, and proxy efficacy with activities such as snack preparation sessions, role-playing games, fruit and vegetable tasting, and playing games that promoted healthier dietary behaviors.
  Interventions: Behavioral: Behavioral nutrition education

INTERVENTIONS:
Behavioral: Behavioral nutrition education — Education aimed at improving knowledge, attitudes, and practices related to dietary intake, with a focus on impacting theorized mediators of nutrition-related behavior.

SUMMARY:
Healthful eating is a core component of a healthy lifestyle that is associated with lower risk of obesity and chronic disease. Although adolescent health promotion programs have been extensively evaluated and applied in English-speaking Western developed nations, there is very little published literature in the Russian context. Our study seeks to determine the relative effectiveness of a healthy lifestyle intervention consisting of nutrition education at a Russian camp. Investigators will determine the impact of behaviorally focused nutrition education on nutrition knowledge, food choice, attitude, and self-efficacy for healthful eating, compared to standard nutrition education.

DETAILED DESCRIPTION:
The project consists of the evaluation of two evidence-based nutrition education programs.

Setting and participants: A random selection of all youth with parental consent for the program will comprise the sample of 40 boys and girls, ages 8-12y. Children with food allergies (to fruits, vegetables, nuts, crackers, corn pops, cookies) will be ineligible for participation. Participants will be randomly assigned to either behaviorally oriented nutrition education or standard nutrition education group (comparison group). Measures: Questionnaires will be completed by each participant at the baseline (the first day) and post-intervention (the last session day). The questionnaire addresses nutrition knowledge, self-efficacy and enjoyment of fruit and vegetable consumption. Controlled observation of healthy/unhealthy snack selection: at the baseline and post-intervention, kids will select snacks first from a menu (individual measure) and then a buffet (group measure) with 3 healthy (fruits and vegetables, nuts) and 3 unhealthy (crackers, corn pops, cookies) snack options. Measurements of height, weight, and waist circumference will be taken prior to the first nutrition education session. Demographics: Investigators will obtain information on age, gender, ethnicity, family socioeconomic status, and parental education level via questionnaire. Procedures: Parents will be informed about potential for child to be involved in healthful nutrition and physical activity at camper check-in. After an informed consent is signed, parents/caregivers and the participant will fill out baseline questionnaires. The parent survey will ask about their child's ethnicity, parental education level, and family socioeconomic status.

Each participant will privately have their height, weight, and waist circumference measured prior to start of study. Participants will attend 45 minute sessions from Monday to Friday throughout 3 weeks at the camp. Each session will be held using different modules from the evidence-based HOP'N After School program. The difference in sessions between the intervention and comparison group will be that the intervention group will get both nutrition education and skill-training component during the session (for example, creating a healthy snack, playing games focusing on enjoyment of fruit and vegetable consumption); the control group will not receive the skill-training component, but will get the same nutrition knowledge as the intervention group. Controlled observation snack tests will take place at the beginning and at the end of the program (baseline and post-intervention).

ELIGIBILITY:
Inclusion Criteria:

* Children attending Yantar, a summer camp in the Northwestern part of Russia (Veshniaki village, Cherepovets district, Vologda region),
* Children of parents who provide permission to participate in a research study

Exclusion Criteria:

* Children outside the 8-12y age range
* Children not randomly selected to participate in nutrition education classes for three weeks.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2014-07-28 (Actual); Study Completion 2015-05-15 (Actual)

PRIMARY OUTCOMES:
Healthy eating choices | Change from Baseline at 3 weeks
  Objective selection of two snacks for consumption from a menu of six choices (direct observation)

SECONDARY OUTCOMES:
Nutrition knowledge | Change from Baseline at 3 weeks
  Questionnaire assessing knowledge related to healthy eating
Healthy eating attitudes | Change from Baseline at 3 weeks
  Questionnaire assessing attitudes related to healthy eating
Fruit and vegetable self-efficacy | Change from Baseline at 3 weeks
  Questionnaire assessing self-efficacy related to eating fruits and vegetables
Fruit and vegetable enjoyment | Change from Baseline at 3 weeks
  Questionnaire assessing enjoyment related to eating fruits and vegetables

CONTACTS AND LOCATIONS:
Overall Officials: Richard R Rosenkranz, PhD, Principal Investigator — Kansas State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: preliminary results — http://hdl.handle.net/2097/19148 — Rodicheva master's thesis document with preliminary analyses